CLINICAL TRIAL: NCT00113334
Title: A Phase 1b/2 Study of ABT-510 (Thrombospondin Analogue) in Patients With Advanced Head and Neck Cancer
Brief Title: Study of ABT-510 (Thrombospondin Analogue) in Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-1027
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2009-06-12 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Thrombospondin Analogue; ABT-510; Antiangiogenic agent; Lung; Skin; Thyroid
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Diseases | interventions — NAc-Sar-Gly-Val-(d-allo-Ile)-Thr-Nva-Ile-Arg-ProNEt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-510 (Thrombospondin) (Experimental): Fixed dose level of thrombospondin 100 mg subcutaneously twice daily.
  Interventions: Drug: ABT-510

INTERVENTIONS:
Drug: ABT-510 — 100 mg subcutaneously twice daily
  Other Names: Thrombospondin Analogue

SUMMARY:
The goals of this clinical research study are to see how individuals with advanced head and neck cancer respond to treatment with the new drug thrombospondin (ABT-510) and to learn how effective it is in destroying cancer cells. The safety of ABT-510 and the effect ABT-510 has on cells in the body will also be studied.

DETAILED DESCRIPTION:
This is a phase Ib/II, single-center, open-label study designed to assess the safety, tolerability, pharmacokinetics, and biologic efficacy of ABT-510 (thrombospondin). Participants will be patients with incurable head and neck cancer.

Patients will begin at a fixed dose level of thrombospondin subcutaneously twice daily. Cycles of treatment are 28 days (4 weeks). Patients will be treated with thrombospondin until progression of tumor or toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically proven squamous cell carcinoma of the head and neck that is not amenable to curative therapy, including radiation or surgery (including surgery following induction chemotherapy or chemo-radiation).
* Patient's tumor is biopsy accessible.
* Patient has a Karnofsky performance status >/= 70.
* Patient has adequate bone marrow function: White blood count (WBC) >/= 3,000 cells/mm3, absolute neutrophil count (ANC) >/= 1,500 cells/mm3, platelet count >/= 100,000 cells/mm3, Hgb >/= 9.0 g/dL.
* Patient has adequate liver function: total bilirubin level </= 2.0 mg/dL, albumin >/= 2.5 g/dL.
* Transaminases (SGOT and/or SGPT) may be up to 2.5 * upper limit of normal (ULN) if alkaline phosphatase is </= ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are </= ULN. However, patients who have both transaminase elevation > 1.5 * ULN and alkaline phosphatase > 2.5 * ULN are not eligible for this study.
* Patient has serum creatinine < 2 mg/dl
* Patient has signed a written informed consent.
* Patient may have received any number of prior chemotherapeutic regimens for recurrent or metastatic disease.
* The subject must not be pregnant or breastfeeding. All subjects (male and female) should practice contraception (e.g., barrier, hormonal, intrauterine device [IUD]) or abstain from sexual intercourse while in the study and for up to two months following completion of therapy.
* The subject is able to self-administer or has a caregiver who can reliably administer subcutaneous (SC) injections.
* Patient >/= 18 years of age.

Exclusion Criteria:

* No biopsy accessible tissue.
* Patient has received prior radiation therapy to biopsy site within the past 3 months. (Patient may have received palliative radiation within the past 2 weeks, but not to the biopsy site.)
* Patient exhibits confusion, disorientation, or has a history of major psychiatric illness which may impair patient's understanding of the informed consent.
* Patient requires total parenteral nutrition with lipids.
* Patient has a history of uncontrolled heart disease including congestive heart failure, angina at rest, myocardial infarct in the last 6 months, uncontrolled hypertension with systolic blood pressure (BP) >160 or diastolic BP >90, systolic blood pressure (BP) <90 or symptomatic hypotension, or symptomatic or potentially life-threatening tachycardia, bradycardia or arrhythmia.
* Pregnant women and women who are currently breast-feeding may not participate in this study. All women of childbearing potential must have a negative pregnancy test within 24 hours prior to enrolling in the study.
* Serious infection or other intercurrent illness requiring immediate therapy.
* The subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g., hemoptysis). The subject has a recent history of (within 4 weeks from Study Day 1) or currently exhibits other clinically significant events of bleeding.
* If subject is receiving therapeutic anticoagulation therapy, low dose anticoagulation for catheter prophylaxis will be permitted; PT/PTT must be within normal limits.
* The patient has a history of or currently exhibits central nervous system (CNS) metastasis. Brain magnetic resonance imaging (MRI) within 28 days of enrollment is required to confirm the absence of CNS metastases.
* Patient has received chemotherapy or biologic therapy within 3 weeks of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward S. Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/10/05 through 03/02/07. All participants recruited at University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | ABT-510 (Thrombospondin)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ABT-510 (Thrombospondin)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 59 [43 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate defined as percentage of number of complete response or partial response in total number of participants treated. Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in sum longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): >20% increase in sum LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1/> new lesions; Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD, reference smallest sum LD. Trial conducted by Simon's optimal two-stage design and response rate estimated accordingly. For status of PR or CR, changes in tumor measurements confirmed by repeat assessments performed at 6 weeks, no less than 4 weeks after criteria for response is first met.
Time Frame: Baseline to 6 weeks for PR or CR response assessment (minimal 4 week cycle + assessments). Overall study period 3 years.
Population: Three (3) patients were inevaluable for response.
Measure: Number; unit: participants
Arm/Group | ABT-510 (Thrombospondin)
Number analyzed (Participants) | 3
participants
  No Change/Stable Disease | 2
  Progressive Disease | 1

ADVERSE EVENTS:
Time Frame: 8 weeks, minimally 28 days for treatment cycle (4 weeks).
Arm/Group | ABT-510 (Thrombospondin)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-510 (Thrombospondin) (N=6)
Fatigue (General disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Metabolism and nutrition disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No